CLINICAL TRIAL: NCT06178250
Title: The Role of Placenta, Fetal Liver, Sectional Ductus Venosus Volumes Examined by Three-dimensional Ultrasound in the Second Trimester in Predicting Gestational Diabetes Mellitus and Maternal-fetal Outcomes
Brief Title: Placenta, Fetal Liver, Sectional Ductus Venosus Volumes Examined by Three-dimensional Ultrasound in the Second Trimester
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011-KAEK-25 2021/10-09
Record Dates: First submitted 2023-12-03; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Gestational Diabetes; DUCTUS VENOSUS VOLUME; PLACENTA VOLUME; 3D SONOGRAPHY; FETAL LİVER VOLUME
Keywords: GESTATİONAL DİABETES MELLİTUS; PLACENTA VOLUME; FETAL LİVER VOLUME; DUCTUS VENOSUS VOLUME; 3D SONUGRAPHY
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: 46 pregnant women diagnosed with gestational diabetes mellitus, 93 pregnant women with normal glycemic index
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- placenta, fetal liver, sectional ductus venosus volumes between 24-29 weeks pregnant women (Other): The placenta, fetal liver and ductus venosus volumes of 46 patients diagnosed with GDM and 93 patients without a GDM diagnosis between 24-29 weeks were evaluated with 3D ultrasound.
  Interventions: Other: 3D sonography

INTERVENTIONS:
Other: 3D sonography — Fetal liver, placenta, and ductus venosus were defined in 3 orthogonal multi-plane images in the voluson 4D view vocal program.
  Other Names: 3D volume description

SUMMARY:
Investigators measured the placenta, fetal liver and ductus venosus volumes of pregnant women with GDM diagnosis and normal glycemic indices in the second trimester.Investigators aimed to correlate measurements with maternal/fetal outcomes and evaluate their success in predicting poor obstetric outcomes

DETAILED DESCRIPTION:
GDM screening may not always be possible with OGTT performed in limited weeks of gestation. In addition, mid-trimester ultrasound scanning is done in all pregnancies. Therefore, measurement of placental volume and fetal liver volume may be an alternative method for the diagnosis of GDM. In order to predict GDM in the second trimester, the use of 3D sonography and VOCAL (Virtual Organ Computer Aided Analysis) technology in high-risk pregnant women and their cost-effectiveness rates should be investigated further. Multicenter randomized controlled studies with more patients are needed to be able to say more clearly.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* diagnosed with GDM

Exclusion Criteria:

* multiple pregnancy
* congenital anomalies
* gestational hypertansion
* preeclampsia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Placenta volume in ultrasound | 10 months
  Measured placenta volumes of pregnant women with GDM diagnosis and normal glycemic indices and evaluate their success in predicting poor obstetrics outcomes
Fetal liver volume in ultrasound | 10 months
  Measured fetal liver and ductus venosus volumes of pregnant women with GDM diagnosis and normal glycemic indices and evaluate their success in predicting poor obstetrics outcomes
Ductus venosus volume in ultrasound | 10 months
  Measured ductus venosus volumes of pregnant women with GDM diagnosis and normal glycemic indices and evaluate their success in predicting poor obstetrics outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)